CLINICAL TRIAL: NCT03572855
Title: The Effect of Peak Scoliosis Spinal Bracing System on Gait and Pain Level in Adult Scoliosis Patients
Brief Title: The Effect Spinal Bracing System on Gait in Adult Scoliosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Texas Back Institute (Other)
Collaborators: Aspen Medical Products (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBIRF-Aspen
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scoliosis Brace (Experimental): The Peak Scoliosis Brace designed to alleviate pain in adult patients with chronic pain secondary to scoliosis.
  Interventions: Combination Product: Scoliosis Brace

INTERVENTIONS:
Combination Product: Scoliosis Brace — Brace will be fitted to each subject by a spine orthopedic surgeon before the testing. The subject will wear the fitted brace for 2 months.

SUMMARY:
Degenerative adult scoliosis (ADS) results from age related changes leading to segmental instability, deformity and stenosis. Patients with scoliosis demonstrate an altered gait pattern.Furthermore, scoliosis patients exert 30% more physical effort than healthy subjects to ensure habitual locomotion, and this additional effort requires a reciprocal increase of oxygen consumption. Bracing has been found to reduce pain within a short time in ADS patients. A new brace has recently become available, the Peak™ Scoliosis Brace (Aspen Medical Products), designed to alleviate pain in adult patients with chronic pain secondary to scoliosis. The purpose of this study is to investigate the impact of spinal bracing using Peak™ Scoliosis Brace on pain and lower extremities kinematics of gait.

DETAILED DESCRIPTION:
Degenerative adult scoliosis (ADS) results from age related changes leading to segmental instability, deformity and stenosis. Although the etiology is unclear, degenerative adult scoliosis is associated with progressive and asymmetric degeneration of the disc and facet joints, which typically leads to stenosis. By virtue of the narrowed spinal canal associated with the degeneration these patients frequently develop back pain, as well as leg pain, weakness, and numbness. With an aging population in the USA and an increased attention to quality of life versus cost issues in the current healthcare environment, degenerative adult scoliosis has become a considerable healthcare concern.

Patients with scoliosis demonstrate an altered gait pattern.Such differences include decreased step length and reduced range of motion in the upper and lower extremities asymmetry of trunk rotation and ground reaction force in three-dimensions. Previous research found a decrease in the muscular mechanical work associated with an increase of energy cost and a decrease in the muscular efficiency in a scoliosis population compared to healthy controls. Furthermore, scoliosis patients exert 30% more physical effort than healthy subjects to ensure habitual locomotion, and this additional effort requires a reciprocal increase of oxygen consumption. This altered gait pattern demonstrated by subjects with scoliosis may be due to changes in global postural control strategies caused by pain and the spinal deformity.

Previous research showed that scoliosis patients do not have impaired postural balance when compared to healthy controls, while several others did find an effect of scoliosis on postural balance. This discrepancy in findings may be due to differences in curve characteristics included and their effects on postural balance, curve types (single or double), number of different curve types, location of curves (thoracic and lumbar), and/or Cobb angles.

Bracing has been found to reduce pain within a short time in ADS patients. Custom-made rigid torso braces, similar to those commonly used for children, are sometimes used in ADS patients; however, only anecdotal evidence of their efficacy is available and problems with comfort and compliance are quite frequent. A new brace has recently become available, the Peak™ Scoliosis Brace (Aspen Medical Products), designed to alleviate pain in adult patients with chronic pain secondary to scoliosis. The Peak Scoliosis Brace led to some improvement of pain at 1 month in a group of adult women with scoliosis and chronic low back pain, but the quality of life did not change significantly. This is may be due to the very short follow-up time. The effect of these braces on functional tasks and activities of daily living including walking have not been studied either.

The purpose of this study is to investigate the impact of spinal bracing using Peak™ Scoliosis Brace on pain and lower extremities kinematics of gait.

METHODS Design This study will be a repeated measurement design. This study will be a non-randomized, prospective, concurrent control cohort study of patients with adult degenerative scoliosis who are clinically indicated for brace intervention and will serve as their own controls via their own pre-treatment evaluation. The proposal design is based on highly recommended Bayesian Design along with the Bayesian and Gaussian analysis for such population and sample size.

Sample Thirty candidates with symptomatic ADS will be enrolled. The sample size needed to approach 80% statistical power for differences between conditions was estimated from the literature.17,23,24 An effect size index of f = 0.50 was estimated. For a desired power of 80% (1 - β = 0.80) and desired α = 0.05, the effect size index requires a minimum sample size of 26.

Inclusion/Exclusion Criteria Thirty spinal deformity patients will be enrolled.

Patients will be classified using the adult deformity SRS-Schwab system. Radiographs made prior to brace treatment and at the two pre-defined follow-up points will be measured and recorded for each patient.

Patients will report to the Spine Biomechanics Laboratory in the Texas Back Institute, be educated on the study and will be asked to provide written informed consent after their questions, if any, are answered. They will then be scheduled for a test session in the lab. Each patient will be evaluated on 2 different occasions: first day of bracing, and 2±0.5 months post-bracing. Subjects will be fitted with 22 external reflective markers. These markers will be placed based on those validated and published in the literature. A static trial will be recorded with subjects positioned in a neutral, standing posture to create a reference for defining neutral joint angles. Each subject will perform a series of over-ground gait trials with self-selected speed. On all visits, subjects will walk 10 meters, stepping on three sequenced force platforms. Subjects will perform a series of gait trials until five acceptable trials are obtained. In addition, each subject will perform 2 additional tests: 1. Timed up and go, and 6 minutes' walk test. After completion of functional testing, the brace will be fitted to each subject by a spine orthopedic surgeon before the testing. The subject will wear the fitted brace for at least 45 minutes prior to retesting. The subject will then repeat the functional testing as mentioned above. Total time required for each subject to participate in one session will be approximately 90 minutes.Three-dimensional (3D) kinematic data will be recorded at 120 Hz via a Vicon-Peak system (Vicon Nexus 2.0 Inc.). Ground reaction force (GRF) (AMTI Corp.) data will be recorded simultaneously at 1200 Hz. Spine, pelvis, hip, knee, and ankle kinematics and GRF will be analyzed using a custom MATLAB program.

Clinical Data Collection Prior to each gait evaluation, patients will be asked to complete a visual analog scale (VAS) to assess back and leg pain intensity, the Oswestry Disability Index (ODI, version 2.1.a), a pain drawing to record symptom location. Patients will also complete an SRS-22r, Fear Avoidance Beliefs Questionnaire (FABQ), and Tampa Scale for Kinesiophobia (TSK) to record how their spinal deformity affects them across several physical and psycho-social domains. Long cassette sagittal and coronal radiographs will be collected at first visit before brace fitting to assess the extent of spinal deformity. As previously stated, the deformity will be measured via the SRS/Schwab deformity classification system.The bracing system to be used is the Peak Scoliosis Bracing System (Aspen Medical Product Inc., Irvine, CA).

The data will be analyzed with a repeated measurement two-way ANOVA to determine differences between pre- and post-bracing measurements. A conservative alpha correction will be made within each statistical family using Bonferroni correction for the multiple dependent variables in order to avoid type I error. Data will also be analyzed to determine whether any outcomes from the gait and balance analysis correlate with patient completed assessments (pain scores) based on Pearson's R correlation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30- 75 years and older
2. Clinically diagnosed thoracolumbar and/or lumbo-sacro-pelvic deformity as defined by the SRS/Schwab classification systems as Cobb angle of 25° or greater
3. Able to ambulate without assistance and stand without assistance with their eyes open for a minimum of 10 seconds
4. Able and willing to attend and perform the activities described in the informed consent within the boundaries of the timelines set forth for pre-, and post-treatment follow-up

Exclusion Criteria:

1. History of prior attempt at fusion (successful or not) at the indicated levels, (history of one level fusion is not an exclusion)
2. Major lower extremity surgery or previous injury that may affect gait (a successful total joint replacement is not an exclusion)
3. BMI higher than 35
4. Neurological disorder, diabetic neuropathy or other disease that impairs the patient's ability to ambulate or stand without assistance
5. Major trauma to the pelvis
6. Pregnant or wishing to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Kinematic Variables Change assessed with human motion capture system | Baseline; 45 minutes and 2 moths after bracing
  3-Dimensional Range of Motion (ROM) during the stance and swing phase of the spine, pelvis, hip, knee, ankle, shoulder, and elbow joint angles along with center of mass and head sway and displacement

SECONDARY OUTCOMES:
Spatio-Temporal Variables Change assessed with human motion capture system | Baseline; 45 minutes and 2 moths after bracing
  Walking speed
Patient Self-Reported Outcome Assessments Change - Visual analog scale (VAS) | Baseline; 45 minutes and 2 moths after bracing
  VAS for lower back pain, neck and arm pain, and leg pain. Scale range from 0 (no pain) - 10 (most pain)
Patient Self-Reported Outcome Assessments Change - Oswestry Disability Index (ODI, version 2.1.a). | Baseline; 45 minutes and 2 moths after bracing
  Scale range from 0 (no pain) - 10 (most pain)
Patient Self-Reported Outcome Assessments Change - Scoliosis Research Society (SRS22) | Baseline; 45 minutes and 2 moths after bracing
  The SRS-22 Patient Questionnaire has become the most widely used patient-reported outcome instrument in the clinical evaluation of patients with idiopathic scoliosis.
Patient Self-Reported Outcome Assessments Change - Tampa Scale for Kinesiophobia (TSK). | Baseline; 45 minutes and 2 moths after bracing
  TSK is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement.
Patient Self-Reported Outcome Assessments Change - Fear Avoidance Beliefs Questionnaire (FABQ) | Baseline; 45 minutes and 2 moths after bracing
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability

CONTACTS AND LOCATIONS:
Overall Officials: Ram Haddas, PhD, Principal Investigator — Texas Back Institute
Locations (1):
- Texas Back Institute, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotwal S, Pumberger M, Hughes A, Girardi F. Degenerative scoliosis: a review. HSS J. 2011 Oct;7(3):257-64. doi: 10.1007/s11420-011-9204-5. Epub 2011 Jun 11. PMID 23024623
- [Background] Kotwicki T, Chowanska J, Kinel E, Czaprowski D, Tomaszewski M, Janusz P. Optimal management of idiopathic scoliosis in adolescence. Adolesc Health Med Ther. 2013 Jul 23;4:59-73. doi: 10.2147/AHMT.S32088. eCollection 2013. PMID 24600296
- [Background] Ploumis A, Transfledt EE, Denis F. Degenerative lumbar scoliosis associated with spinal stenosis. Spine J. 2007 Jul-Aug;7(4):428-36. doi: 10.1016/j.spinee.2006.07.015. Epub 2007 Feb 28. PMID 17630141
- [Background] Engsberg JR, Bridwell KH, Reitenbach AK, Uhrich ML, Baldus C, Blanke K, Lenke LG. Preoperative gait comparisons between adults undergoing long spinal deformity fusion surgery (thoracic to L4, L5, or sacrum) and controls. Spine (Phila Pa 1976). 2001 Sep 15;26(18):2020-8. doi: 10.1097/00007632-200109150-00016. PMID 11547203
- [Background] Yang JH, Suh SW, Sung PS, Park WH. Asymmetrical gait in adolescents with idiopathic scoliosis. Eur Spine J. 2013 Nov;22(11):2407-13. doi: 10.1007/s00586-013-2845-y. Epub 2013 Jun 4. PMID 23732766
- [Background] Mahaudens P, Banse X, Mousny M, Detrembleur C. Gait in adolescent idiopathic scoliosis: kinematics and electromyographic analysis. Eur Spine J. 2009 Apr;18(4):512-21. doi: 10.1007/s00586-009-0899-7. Epub 2009 Feb 18. PMID 19224255
- [Background] Arima H, Yamato Y, Hasegawa T, et al. Gait analysis after corrective surgery for adult spinal deformity - good sagittal balance with improved lumber lordosis is important. Scoliosis 2015;10:O76
- [Background] Kramers-de Quervain IA, Muller R, Stacoff A, Grob D, Stussi E. Gait analysis in patients with idiopathic scoliosis. Eur Spine J. 2004 Aug;13(5):449-56. doi: 10.1007/s00586-003-0588-x. Epub 2004 Apr 3. PMID 15064994
- [Background] Schizas CG, Kramers-de Quervain IA, Stussi E, Grob D. Gait asymmetries in patients with idiopathic scoliosis using vertical forces measurement only. Eur Spine J. 1998;7(2):95-8. doi: 10.1007/s005860050037. PMID 9629931
- [Background] Chockalingam N, Dangerfield PH, Rahmatalla A, Ahmed el-N, Cochrane T. Assessment of ground reaction force during scoliotic gait. Eur Spine J. 2004 Dec;13(8):750-4. doi: 10.1007/s00586-004-0762-9. Epub 2004 Jun 22. PMID 15221574
- [Background] Giakas G, Baltzopoulos V, Dangerfield PH, Dorgan JC, Dalmira S. Comparison of gait patterns between healthy and scoliotic patients using time and frequency domain analysis of ground reaction forces. Spine (Phila Pa 1976). 1996 Oct 1;21(19):2235-42. doi: 10.1097/00007632-199610010-00011. PMID 8902968
- [Background] Mahaudens P, Detrembleur C, Mousny M, Banse X. Gait in adolescent idiopathic scoliosis: energy cost analysis. Eur Spine J. 2009 Aug;18(8):1160-8. doi: 10.1007/s00586-009-1002-0. Epub 2009 Apr 24. PMID 19390877
- [Background] O'Beirne J, Goldberg C, Dowling FE, Fogarty EE. Equilibrial dysfunction in scoliosis--cause or effect? J Spinal Disord. 1989 Sep;2(3):184-9. PMID 2520074
- [Background] Kuo FC, Wang NH, Hong CZ. Impact of visual and somatosensory deprivation on dynamic balance in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2010 Nov 1;35(23):2084-90. doi: 10.1097/BRS.0b013e3181cc8108. PMID 20975488
- [Background] Karimi MT, Kavyani M, Kamali M. Balance and gait performance of scoliotic subjects: A review of the literature. J Back Musculoskelet Rehabil. 2016 Aug 10;29(3):403-15. doi: 10.3233/BMR-150641. PMID 26519115
- [Background] Beaulieu M, Toulotte C, Gatto L, Rivard CH, Teasdale N, Simoneau M, Allard P. Postural imbalance in non-treated adolescent idiopathic scoliosis at different periods of progression. Eur Spine J. 2009 Jan;18(1):38-44. doi: 10.1007/s00586-008-0831-6. Epub 2008 Dec 6. PMID 19066989
- [Background] Schimmel JJ, Groen BE, Weerdesteyn V, de Kleuver M. Adolescent idiopathic scoliosis and spinal fusion do not substantially impact on postural balance. Scoliosis. 2015 Jun 9;10:18. doi: 10.1186/s13013-015-0042-y. eCollection 2015. PMID 26056528
- [Background] Guo X, Chau WW, Hui-Chan CW, Cheung CS, Tsang WW, Cheng JC. Balance control in adolescents with idiopathic scoliosis and disturbed somatosensory function. Spine (Phila Pa 1976). 2006 Jun 15;31(14):E437-40. doi: 10.1097/01.brs.0000222048.47010.bf. PMID 16778672
- [Background] Simoneau M, Mercier P, Blouin J, Allard P, Teasdale N. Altered sensory-weighting mechanisms is observed in adolescents with idiopathic scoliosis. BMC Neurosci. 2006 Oct 19;7:68. doi: 10.1186/1471-2202-7-68. PMID 17052338
- [Background] Marcotte L. SpineCor in the treatment of adult. Scoliosis 2010;5:47.
- [Background] Zaina F, Poggio M, Donzelli S, Negrini S. Can bracing help adults with chronic back pain and scoliosis? Short-term results from a pilot study. Prosthet Orthot Int. 2018 Aug;42(4):410-414. doi: 10.1177/0309364618757769. Epub 2018 Feb 15. PMID 29446692
- [Background] Gallo D. Case reports: orthotic treatment of adult scoliosis patients with chronic back pain. Scoliosis. 2014 Nov 18;9:18. doi: 10.1186/1748-7161-9-18. eCollection 2014. PMID 25904972
- [Background] Sachs D, Capobianco R, Cher D, Holt T, Gundanna M, Graven T, Shamie AN, Cummings J Jr. One-year outcomes after minimally invasive sacroiliac joint fusion with a series of triangular implants: a multicenter, patient-level analysis. Med Devices (Auckl). 2014 Aug 28;7:299-304. doi: 10.2147/MDER.S56491. eCollection 2014. PMID 25210479
- [Background] Toosizadeh N, Yen TC, Howe C, Dohm M, Mohler J, Najafi B. Gait behaviors as an objective surgical outcome in low back disorders: A systematic review. Clin Biomech (Bristol). 2015 Jul;30(6):528-36. doi: 10.1016/j.clinbiomech.2015.04.005. Epub 2015 Apr 17. PMID 25921552
- [Background] Portney LG, Watkins MP. Foundation of clinical research: applications to practice. 3rd ed. Upper Saddle River, New Jersy: Julie Levin Alexander, 2009.
- [Background] Sengupta DK. Re: Schwab F, Ungar B, Blondel B, et al. Scoliosis research society-Schwab adult spinal deformity classification--a validation study. Spine 2012; 37:1077-82. Spine (Phila Pa 1976). 2012 Sep 15;37(20):1790. doi: 10.1097/BRS.0b013e318260d8e4. No abstract available. PMID 22976199
- [Background] El Fegoun AB, Schwab F, Gamez L, Champain N, Skalli W, Farcy JP. Center of gravity and radiographic posture analysis: a preliminary review of adult volunteers and adult patients affected by scoliosis. Spine (Phila Pa 1976). 2005 Jul 1;30(13):1535-40. doi: 10.1097/01.brs.0000167534.49069.e9. PMID 15990669
- [Background] Vaughan CL, Davis BL, O'Conner JC. Dynamics of Human Gait. 2nd ed. Cape Town, South Africa: Kiboho Publishers, 1999.